CLINICAL TRIAL: NCT02980861
Title: Laparoscopic Versus Open Total Gastrectomy With Spleen-preserving Splenic Hilum Lymph Nodes Dissection for Advanced Proximal Gastric Cancer: A Randomized Controlled Trial
Brief Title: Laparoscopic Versus Open Gastrectomy With Splenic Hilum Lymph Nodes Dissection
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Lin Chen, Director, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Z161100000516237
Record Dates: First submitted 2016-11-30; First posted 2016-12-02 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer; Splenic Hilum Lymph Nodes Dissection; Gastrectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopic total gastrectomy (Experimental): Participants including in the laparoscopic total gastrectomy (LTG) group will undergo LTG with spleen-preserving splenic hilum lymph nodes dissection.
  Interventions: Procedure: Laparoscopic total gastrectomy
- Open total gastrectomy (Active Comparator): Participants who are included in the open total gastrectomy (OTG) group will OTG with spleen-preserving splenic hilum lymph nodes dissection.
  Interventions: Procedure: Open total gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic total gastrectomy — When the participants with advanced proximal gastric cancer are randomized in the laparoscopic totalgastrectomy (LATG) group, they will received LTG with spleen-preserving splenic hilum lymph nodes dissection.
  Other Names: LTG
  Arms: Laparoscopic total gastrectomy
Procedure: Open total gastrectomy — When the participants with advanced proximal gastric cancer are randomized in the open total gastrectomy(OTG) group, they will received OTG with spleen-preserving splenic hilum lymph nodes dissection.
  Other Names: OTG
  Arms: Open total gastrectomy

SUMMARY:
Splenic hilum remains challenging during total gastrectomy with D2 lymphadenectomy.The application of minimally invasive surgery for advanced gastric cancer is gaining popularity. The investigators aim to compare the safety and feasibility of LTG and OTG for advanced proximal gastric cancer.

DETAILED DESCRIPTION:
Total gastrectomy with D2 lymphadenectomy remains the standard surgical therapy for patients with advanced proximal gastric cancer. Although lymph nodes dissection along with the splenic hilum (No.10) is recommended by the Japanese Gastric Cancer Treatment Guidelines, however, complete removal of the No. 10 is technically challenging due to the tortuous splenic vessels and the high possibility of injury to the parenchyma of the spleen and pancreas. Recently, the application of minimally invasive surgery for advanced gastric cancer is gaining popularity. However, laparoscopic total gastrectomy (LTG) with standard D2 lymphadenectomy was still not widely performed, because pancreas- and spleen-preserving splenic hilum lymph node dissection were mainly challenging manipulations for laparoscopic surgeons. Therefore,the investigators aim to investigate the safety and feasibility of LTG with spleen-preserving splenic hilum lymph node dissection for proximal advanced gastric cancer and compare the early results of this procedure with open total gastrectomy (OTG).

ELIGIBILITY:
Inclusion Criteria:

1. Primary proximal gastric adenocarcinoma confirmed pathologically by endoscopic biopsy;
2. cT2-4aN0-3M0 at preoperative evaluation according to American Joint Committee On Cancer (AJCC) Cancer Staging Manual, 7th Edition.
3. Eastern Cooperative Oncology Group (ECOG): 0 or 1;
4. American Society of Anesthesiologists （ASA） score: Ⅰto Ⅲ;
5. Written informed consent.

Exclusion Criteria:

1. Pregnant or breast-feeding women;
2. Severe mental disorder;
3. Previous upper abdominal surgery (except laparoscopic cholecystectomy);
4. Previous gastrectomy, endoscopic mucosal resection, or endoscopic submucosal dissection;
5. Enlarged or bulky regional lymph node diameter larger than 3 cm based on preoperative imaging;
6. Other malignant disease within the past 5 years;
7. Previous neoadjuvant chemotherapy or radiotherapy;
8. Contraindication to general anesthesia (severe cardiac and/or pulmonary disease);
9. Emergency surgery due to a complication (bleeding, obstruction, or perforation) caused by gastric cancer.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Number of group Splenic Hilum (No.10) lymph nodes harvested | 7 days

SECONDARY OUTCOMES:
Early complication rate | 30 days
  The early complication rate is defined as the event observed during operation
Operative time | Intraoperative
Operative blood loss | Intraoperative
Time of splenic hilum lymph nodes dissection | Intraoperative
Number of total lymph nodes harvested | 7 days
Post-operative recovery course | 30 days
  Time to first ambulation, flatus, liquid diet and duration of hospital stay are used to assess the postoperative recovery course
3-year disease free survival rate | 3 years
3-year overall survival rate | 3 years
Quality of life | 1 year
  It will be assessed by questionnaire (WHO quality of life-100)

CONTACTS AND LOCATIONS:
Overall Officials: Lin Chen, Principal Investigator — the Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bian S, Xi H, Wu X, Cui J, Ma L, Chen R, Wei B, Chen L. The Role of No. 10 Lymphadenectomy for Advanced Proximal Gastric Cancer Patients Without Metastasis to No. 4sa and No. 4sb Lymph Nodes. J Gastrointest Surg. 2016 Jul;20(7):1295-304. doi: 10.1007/s11605-016-3113-3. Epub 2016 Mar 3. PMID 26940944
- [Derived] Guo X, Peng Z, Lv X, Cui J, Zhang K, Li J, Jin N, Xi H, Wei B, Chen L. Randomized controlled trial comparing short-term outcomes of laparoscopic and open spleen-preserving splenic hilar lymphadenectomy for advanced proximal gastric cancer: An interim report. J Surg Oncol. 2018 Dec;118(8):1264-1270. doi: 10.1002/jso.25262. Epub 2018 Oct 31. PMID 30380145